CLINICAL TRIAL: NCT06488157
Title: Adapting and Implementing the I-HoME Intervention in Caregivers of Patients With ADRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-01025643; K76AG059997-04S1 (NIH)
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (I-HoME) (Experimental): Participants receive video visits with a nurse practitioner for up to six visits every 2 weeks to address symptom management and care needs.
  Interventions: Other: I-HoME

INTERVENTIONS:
Other: I-HoME — Video visits with a nurse practitioner for up to six visits every 2 weeks to address symptom management and care needs

SUMMARY:
The purpose of this study is to pilot test the adapted Improving Home hospice Management of End-of-life issues through technology (I-HoME) intervention with family caregivers of patients with advanced Alzheimer's Disease and related dementia. Data will be collected regarding intervention feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and < 100 years
* English speaking
* Providing care to an ADRD patient who is age ≥ 65 years old and < 105 years who is a stage 7a-f on the Functional Assessment Staging Tool (FAST) scale

Exclusion Criteria:

* Non-English speaking
* <18 years old or >100 years old

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veerawat Phongtankuel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention (I-HoME)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention (I-HoME)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Highest Education Completed [Count of Participants; unit: Participants]
  Some high school | 0
  High School or GED | 0
  Some College | 2
  College degree | 1
  Post-graduate but no degree | 0
  Graduate Degree | 12
Annual Household Income Range [Count of Participants; unit: Participants]
  $25,000 or less | 0
  $25,001 to $50,000 | 1
  $50,001 to $75,000 | 2
  $75,001 or greater | 12
Relationship to Patient [Count of Participants; unit: Participants]
  Spouse/partner | 4
  Child | 10
  Relative | 1
  Friend | 0
  Paid Caregiver | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility, as Measured by the Percentage of Caregivers Who Enroll in the Study
Description: Feasibility was measured by the percentage of caregivers who enrolled in the study out of all eligible participants.
Time Frame: Recruitment (7 months)
Population: All participants who we reached out to and were eligible for our study, including those who refused to participate or were unreachable over multiple attempts, were included in the number of participants analyzed for this measure.
Measure: Number; unit: percentage of all eligible participants
Groups:
- All Participants: This measure represents the recruitment rate for all participants.
Arm/Group | All Participants
Number analyzed (Participants) | 41
percentage of all eligible participants | 37

2. Primary Outcome: Feasibility, as Measured by the Percentage of Tele-visits Conducted
Description: Feasibility was measured by dividing the number of tele-visits conducted by the number of tele-visits that could have been conducted, then multiplying by 100. This measure shows the adherence of the intervention arm to the tele-visits. The percentage is calculated for the group rather than the individual patient.
Time Frame: At the end of the intervention or at 12 weeks, whichever is earlier
Measure: Number; unit: percentage of tele-visits conducted
Units Other Than Participants: Tele-visits
Arm/Group | Intervention (I-HoME)
Number analyzed (Participants) | 15
Number analyzed (Tele-visits) | 90
percentage of tele-visits conducted | 95.5

3. Secondary Outcome: Change in Behavioral and Psychosocial Symptoms of Dementia (BPSD) in the Patient, as Measured by the Neuropsychiatric Inventory Questionnaire
Description: Change in behavioral and psychosocial symptoms of dementia (BPSD) in the patient, as measured by the Neuropsychiatric Inventory Questionnaire. Scale is from 0 to 36, with higher scores indicating more severe BPSD.
Time Frame: Baseline, 2, 4, 6, 8, 10, 12 weeks
Population: This measure was not collected because, after completing the first phase of the study, we found it was not relevant to the participants in the clinical trial.
Arm/Group | Intervention (I-HoME)
Number analyzed (Participants) | 0

4. Secondary Outcome: Mean Caregiver Depression Score, as Measured by Patient Health Questionnaire-8
Description: Mean caregiver depression score, as measured by Patient Health Questionnaire-8. Scale is from 0 to 24, with higher scores indicating more severe depression.
Time Frame: Baseline, 2, 4, 6, 8, 10, 12 week
Population: The number of participants analyzed at each time point varied because:
  A caregiver was ineligible to participate due to their care recipient passing away.
  A caregiver missed the tele-visit session on that particular week.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (I-HoME)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 4.8 (3.03)
  Week 2 | 4.5 (2.77)
  Week 4: number analyzed (Participants) | 14
  Week 4 | 3.3 (2.70)
  Week 6 | 3.4 (3.38)
  Week 8: number analyzed (Participants) | 14
  Week 8 | 3.6 (3.15)
  Week 10: number analyzed (Participants) | 14
  Week 10 | 4.5 (3.74)
  Week 12 | 3.5 (2.10)

5. Secondary Outcome: Mean Caregiver Anxiety Score, as Measured by General Anxiety Disorder-7
Description: Mean caregiver anxiety score, as measured by General Anxiety Disorder-7. Scale is from 0 to 21, with higher scores indicating more severe anxiety.
Time Frame: Baseline, 2, 4, 6, 8, 10, 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (I-HoME)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 5.9 (3.25)
  Week 2 | 5.0 (4.17)
  Week 4: number analyzed (Participants) | 14
  Week 4 | 4.3 (3.77)
  Week 6 | 3.9 (3.96)
  Week 8: number analyzed (Participants) | 14
  Week 8 | 4.7 (4.94)
  Week 10: number analyzed (Participants) | 14
  Week 10 | 5.0 (4.49)
  Week 12 | 3.4 (3.33)

6. Secondary Outcome: Mean Caregiver Burden Score, as Measured by the Zarit Burden Interview - Short Version
Description: Mean caregiver burden score, as measured by the Zarit Burden Interview - short version. Scale is from 0 to 48, with higher scores indicating higher caregiver burden.
Time Frame: Baseline, 2, 4, 6, 8, 10, 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (I-HoME)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 16.6 (6.54)
  Week 2 | 12.1 (7.43)
  Week 4: number analyzed (Participants) | 14
  Week 4 | 10.1 (5.90)
  Week 6 | 9.7 (6.17)
  Week 8: number analyzed (Participants) | 14
  Week 8 | 9.6 (7.02)
  Week 10: number analyzed (Participants) | 14
  Week 10 | 10.6 (6.33)
  Week 12 | 10.6 (7.00)

7. Secondary Outcome: Mean Caregiver Perception of Patient's Pain Score, as Measured by the Doloplus 2 Scale Behavioral Assessment
Description: Mean caregiver perception of patient's pain score, as measured by the Doloplus 2 Scale behavioral assessment. Scale is from 0 to 30, with higher scores indicating greater pain.
Time Frame: Baseline, 2, 4, 6, 8, 10, 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (I-HoME)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 5.1 (3.99)
  Week 2 | 3.9 (2.83)
  Week 4: number analyzed (Participants) | 14
  Week 4 | 3.7 (2.49)
  Week 6 | 3.5 (4.02)
  Week 8: number analyzed (Participants) | 14
  Week 8 | 3.4 (3.92)
  Week 10: number analyzed (Participants) | 14
  Week 10 | 4.4 (4.62)
  Week 12 | 4.1 (4.08)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Only caregivers of patients with ADRD, not their care recipients, were assessed for adverse events.
Arm/Group | Intervention (I-HoME)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT06488157/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT06488157/ICF_001.pdf